CLINICAL TRIAL: NCT02271308
Title: The Effects of Low Resistance Training Using Elastic Band on Muscle Strength, Flexibility, Quality of Life and Ease of Care in Nursing Home Residents: A Pilot Study
Brief Title: The Effects of Low Resistance Training on the Residents in Nursing Homes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chang Bing Show Chwan Memorial Hospital (Other)
Responsible Party: Principal Investigator, Shu-Hui Yeh, RN, PhD, Professor, Chang Bing Show Chwan Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 1030109
Record Dates: First submitted 2014-10-14; First posted 2014-10-22 (Estimated); Last update posted 2014-10-22 (Estimated); Status verified 2014-10

CONDITIONS: Elderly Residents
Keywords: elastic band resistance training; nursing home residents; muscle strength; flexibility; quality of life; ease of care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control group (No Intervention): Residents in control group will receive regular activity in nursing homes.
- Experimental group (Experimental): The residents in experimental group will receive a low-resistance elastic band training (30 minutes), including warm-up and cold-down period, three times per week for 12 weeks.
  Interventions: Behavioral: Low-resistance elastic band training

INTERVENTIONS:
Behavioral: Low-resistance elastic band training — The residents in experimental group will receive a low-resistance elastic band training (30 minutes), including warm-up and cold-down period, three times per week for 12 weeks.
  Arms: Experimental group

SUMMARY:
This study will examine the effects of low-resistance elastic band training on muscle strength, flexibility, quality of life and ease of care among the residents in nursing homes.

DETAILED DESCRIPTION:
Regular exercise and dynamic life style can prevent and treat disability, as well as promote mental health and quality of life. In addition to chronic illness, reduced muscle mass and strength as part of aging, affect the daily activities of living of the elderly and their independent lifestyle. In fact, exercise had found positive effects on lower limb weakness of the elderly. Elastic band is a resistance training aid which can be used for different muscle weight training. The research results have been demonstrated elastic band resistance training is safe and effective strategy to apply in the elderly population and to improve physical fitness, and mental functioning. Therefore, this study will examine the effects of low-resistance elastic band training on muscle strength, flexibility, quality of life and ease of care among the nursing home residents. Nursing homes with more than 50 beds that will be recruited in Qingshui and Waipu district Taichung City. Nursing homes will be randomly assigned to the experimental group and the comparison group. Each group has 20 subjects. The residents in experimental group will receive a low-resistance elastic band training(30 minutes), including warm-up and cold-down period, three times per week for 10 weeks. Residents in control group will receive regular activity in nursing home. Inclusion criteria for the elderly include: (1) living in nursing home over 3 months; (2) communicating with Mandarin and Taiwanese; (3) being able to sit in a chair or wheelchair; (4) can grip elastic band by hands; (5) no severe cardiovascular disease, musculoskeletal disorders and mental illness;(6) consciousness intact and their consent to participate in this study. Two structured questionnaires and an assessment checklist of muscle strength, flexibility will be used to collect data at baseline, week 8 and week 12 of exercise. The collected data will be coded and double checked and analyzed by using SPSS Window Release 20.0. The findings of this study can be apply to develop and conduct an effective exercise program through elastic band resistance training to improve residents' strength, flexibility, quality of life and care of ease in Taiwan.

ELIGIBILITY:
Inclusion Criteria:

* living in nursing home over 3 months
* communicating with Mandarin and Taiwanese
* being able to sit in a chair or wheelchair
* can grip elastic band by hands
* consciousness intact and their consent to participate in this study

Exclusion Criteria:

* severe cardiovascular disease, musculoskeletal disorders and mental illness

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2014-03; Primary Completion 2015-02 (Estimated); Study Completion 2015-02 (Estimated)

PRIMARY OUTCOMES:
Improve muscle strength | Change from baseline in muscle strength at 3 months
  Muscle strength will be assessed using hand-held dynameter at 3 different times: (1) baseline data: before low-resistance elastic band training, (2) outcome data: at 8 and 12 weeks post-test.

SECONDARY OUTCOMES:
Improve body flexibility | Change from baseline in Body flexibility at 3 months
  Body flexibility will be assessed at 3 different times: (1) baseline data: before low-resistance elastic band training, (2) outcome data: at 8 and 12 weeks post-test.
Improve life quality | Change from baseline in life quality at 3 months
  Life quality will be assessed by SF-12 questionnaire（Short Form-12 Items Health Survey,SF-12）at 3 different times: (1) baseline data: before low-resistance elastic band training, (2) outcome data: at 8 and 12 weeks post-test.
Improve quality of care | Change from baseline in quality of care at 3 months
  Quality of care will be assessed by ease-of-care inventory (Yan、Wu、 Lin and Lin, 2007) at at three different times: (1) baseline data :before low-resistance elastic band training, (2) outcome data: at 8 and 12 weeks post-test.
Basic attribute data | Change from baseline in basic attribute data at 3 months
  Subjects will fill out questionnaire including blood pressure, pulse, activity, respiration, pain, ADL (Barthel Index), weight, thickness of subcutaneous fat and body mass index (BMI).

CONTACTS AND LOCATIONS:
Overall Officials: Li-Wei Lin, PhD., Principal Investigator — Department of Nursing, Hung Kuang University; Shu-Hui Yeh, PhD., Principal Investigator — Chang Bing Show Chwan Memorial Hospital & Central Taiwan University of Science and Technology
Locations (1):
- Division of Core Laboratory; Chang Bing Show Chwan Memorial Hospital, Changhua County, Taiwan